CLINICAL TRIAL: NCT04586218
Title: Postoperative Hypotension Management With Computer-guided Vasopressor Titration in High-Risk Patients After Cardiac Surgery: A Randomized Controlled Trial
Brief Title: Controling Mean Arterial Pressure Using a Closed-Loop System for Vasopressor Titration
Acronym: COMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique de la Sauvegarde (Other)
Collaborators: Bicetre Hospital (Other); Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019-A03191-56
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Intervention Model Description: Randomized controlled superiority trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual control of vasopressor infusion (Active Comparator): Vasopressor will be manually titrated by intensive care unit nurses in charge of the patients to maintain mean arterial pressure > 65 mmHg.
  Fluid administration consists in optimization of stroke volume (assisted fluid management) during the postoperative period
  Interventions: Behavioral: Manual control of vasopressor infusion
- Computer guided vasopressor infusion (Experimental): Vasopressor will be titrated automatically by the closed-loop system to maintain mean arterial pressure > 65 mmHg.
  Fluid administration consists in optimization of stroke volume (assisted fluid management) during the postoperative period
  Interventions: Behavioral: Computer guided vasopressor infusion

INTERVENTIONS:
Behavioral: Computer guided vasopressor infusion — automated titration of vasopressor infusion to maintain a mean arterial pressure > 65mmHg
  Arms: Computer guided vasopressor infusion
Behavioral: Manual control of vasopressor infusion — manual adjustments of noradrenaline infusion
  Arms: Manual control of vasopressor infusion

SUMMARY:
The investigators have developed an automated vasopressor controller to improve the titration of vasopressor in order to maintain mean arterial pressure (MAP) within a narrow range and have recently shown the controller was effective in both the operating room and intensive care unit. The controller has been used recently in a case series of three patients undergoing cardiac surgery and in five patients after cardiac surgery.

The investigators want to compare now a manual to a closed-loop titration of vasopressor infusion in patients admitted in the Intensive Care unit after cardiac surgery

DETAILED DESCRIPTION:
Perioperative hypotension and arterial pressure variability have been shown to negatively impact patient outcomes, increasing risk of stroke, kidney injury, and myocardial injury among others.

Vasopressors are usually used to rapidly correct hypotension. Vasopressor infusions are typically administered by standard infusion pump with the rate adjusted by anesthesiologists to reach a predefined target mean arterial pressure (MAP); this requires frequent changes in the infusion rate because of the almost constantly changing hemodynamic status of such patients. Because it is infeasible for human providers to pay constant attention and make second-to-second changes, management is often suboptimal (i.e. large amounts of time are spent in hypotension below the target, or well above the target with the vasopressor drip still running).

The investigators have developed an automated closed-loop vasopressor (CLV) controller to improve the titration of vasopressor (e.g:noradrenaline) in order to maintain MAP within a narrow range in the perioperative setting. The investigators have published engineering, animal and most recently, pilot,studies or case series with promising results.

In this randomized controlled trial, the investigators will compare time spent in hypotension defined as a mean arterial pressure < 65 mmHg. They tested the hypothesis that the automated system will allow patients to spent less time during the postoperative period with a MAP < 65 mmHg. This is thus a superiority study over a two hours study period

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Elective cardiac surgery
* French speaking patient

Exclusion Criteria:

* Uncontrolled hypertension
* Renal insufficiency (estimated glomerular filtration rate < 30mL/min/1,73m²)
* Left ejection fraction < 40%
* Emergency surgery
* Preoperative infection
* Preoperative cardiac arrythmia
* Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative hypotension | postoperative hour 2
  Percentage of treatment period spent with a MAP < 65 mmHg

SECONDARY OUTCOMES:
Number of vasopressor infusion rate modifications | postoperative hour 2
  Number of vasopressor infusion rate modifications
Amount of vasopressor | postoperative hour 2
  Amount of noradrenaline received during surgery
amount of fluid | postoperative hour 2
  amount of fluid received during surgery
incidence of acute kidney injury | postoperative day 7
  incidence of acute kidney injury at postoperative day 7
troponin values | postoperative day 0
  troponin values at intensive care arrival
troponin values | postoperative day 1
  troponin values at postoperative day 1

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Desebbe, MD, Principal Investigator — Clinique de la Sauvegarde
Locations (1):
- Clinique de la Sauvegarde, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desebbe O, Rinehart J, Van der Linden P, Cannesson M, Delannoy B, Vigneron M, Curtil A, Hautin E, Vincent JL, Duranteau J, Joosten A. Control of Postoperative Hypotension Using a Closed-Loop System for Norepinephrine Infusion in Patients After Cardiac Surgery: A Randomized Trial. Anesth Analg. 2022 May 1;134(5):964-973. doi: 10.1213/ANE.0000000000005888. PMID 35061635